CLINICAL TRIAL: NCT05669131
Title: Motor Imagery Training, Force Steadiness and Neural Drive
Brief Title: Does Motor Imagery Training Enhance Control of Movement in Older Adults?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Jakobi, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MIT&ForceSteadiness
Record Dates: First submitted 2022-11-29; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Aged; Aged, 80 and over

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the motor imagery training group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery Training (Experimental): Participants will do motor imagery training in 5 minute blocks for a total of 20 minutes.
  Interventions: Other: Motor imagery training
- Control (No Intervention): Participants will watch a documentary in 5 minute blocks for a total of 20 minutes.

INTERVENTIONS:
Other: Motor imagery training — Participants imagine themselves through their own eyes performing submaximal elbow flexion contractions.
  Arms: Motor Imagery Training

SUMMARY:
The goal of this clinical trial is learn about motor imagery training (i.e. imagining a task) with healthy older adults. The main question this clinical trial aims to answer is:

• Will imagining a task improve control of force during an elbow flexion muscle contraction in healthy older adults?

Participants will:

* Complete questionaries about general activity levels and ability to imagine tasks
* Perform either motor imagery training or watch a documentary
* Perform maximal and submaximal elbow flexion contractions

Researchers will compare the motor imagery training with the control group to see if control of force is improved in the motor imagery training group.

DETAILED DESCRIPTION:
Motor imagery training could be beneficial in rehabilitative settings when participants are not physically capable of preforming a motor task or in injury prevention scenarios such as when multiple repetitions of a motor task should not be performed. If the effects of motor imagery training are favourable then they could have meaningful influence on the performance of steady movements in older adults who experience declines in force steadiness with age. Therefore, the first aim of this study will be to determine if one session of motor imagery training will influence corticospinal excitability in older adults and improve force steadiness during isometric elbow flexion contractions with the observed benefit being greater in females. The second aim of this study will be to determine if there is an associated change in oscillations in common synaptic input to motor neurons with a change in force steadiness.

ELIGIBILITY:
Inclusion Criteria:

Healthy older adults aged 65 to 90 years old

Exclusion Criteria:

1. have had an injury or orthopaedic surgery to the arm or shoulder in the prior 6 months
2. are involved in high levels of upper-body strength training
3. have history of training in fine motor tasks (i.e., musicians)
4. have a history of MIT
5. have systemic diseases and/or nerve damage affecting neuromuscular function
6. have severe cognitive impairment
7. are unable to read or speak English fluently
8. are left hand dominant

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Force steadiness | Within one session: Change from baseline (immediately before session) to 20 minutes after the session
  Measured as the the coefficient in variation of force
Corticospinal excitability | Within one session: Change from baseline (immediately before session) to 20 minutes after the session
  Measured as the peak-to-peak amplitude of a motor evoked potential
Common synaptic input | Within one session: Change from baseline (immediately before session) to 20 minutes after the session
  Estimated from motor unit discharge times.

SECONDARY OUTCOMES:
Maximal elbow flexion force | Within one session: Change from baseline (immediately before session) to 20 minutes after the session
  The total amount of force produced during a maximal contraction

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jakobi, PhD, Principal Investigator — University of British Columbia- Okanagan